CLINICAL TRIAL: NCT01401972
Title: Conventional and Contrast-Assisted Frequency Functional Ultrasound for Imaging of Prostate Cancer Extent and Response in Human Cancer Patients
Brief Title: Conventional Ultrasound for Imaging of Prostate Cancer Extent and Response in Human Cancer Patients
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Dr., Sunnybrook Health Sciences Centre
Other Study IDs: Ultrasound Prostate Cancer
Record Dates: First submitted 2010-09-01; First posted 2011-07-26 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; ultrasound; spectroscopy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Prostate speciments are retained after radical prostatectomy surgery
Oversight: Data Monitoring Committee: No

SUMMARY:
In this observational study the investigators will undertake imaging studies on men with prostate cancer. The primary hypothesis is that ultrasound spectroscopy could be used to determine the extent of disease inside and outside of the prostate gland in patients with prostate cancer. It is hoped that the changes in ultrasound backscatter parameters obtained before radical prostatectomy could be used to correlate with pathological findings from the prostate specimen after surgery.

DETAILED DESCRIPTION:
This project is an early validation study in human subjects that will use ultrasound imaging and spectroscopy to predict the tumour extent before treatment so that this may allow the most appropriate treatment intervention to be individualised to patients. For examples, patients with evidence of extra-prostatic tissue involvement may be best served with definitive radiation therapy rather than radical prostatectomy as surgery alone in this situation, is not optimum. Furthermore, these ultrasound parameters may be used to monitor cell death occurring at various time points during patients' radiation treatment for prostate cancer.

The research is exploratory since upon data analysis it will examine the use of different ultrasound parameters as potential markers of pre-treatment tumour extent and cell death, and correlate these with tumour shrinkage and complete pathological response. Sensitivity and specificity values for the various ultrasound parameters will be calculated for the different time points used and receiver-operator curves will be generated. From this data the investigators will potentially estimate the best time-points at which to make a prediction about patient response and the best ultrasound-spectroscopy variables to use for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Prostate Cancer

Exclusion Criteria:

* Not having radical prostatectomy surgery

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will investigate a population of 30 men with prostate cancer undergoing radical prostatectomy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
ultrasound backscatter parameters such as aggregate mid-band fit, spectroscopic slope and intercept and the number of vessels with detectable blood flow and their sizes | Up to year 2019
  These parameters will be obtained before radical prostatectomy to correlate with pathological findings from the prostate specimen after surgery.

SECONDARY OUTCOMES:
sensitivity and specificity of ultrasound-based imaging of the prostate | Up to year 2019
  the changes in the ultrasound backscatter parameters obtained from the ultrasonic spectroscopy during patient's radiation treatment would be used to monitor tumor response and to correlate with pathological findings in patients with prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Czarnota, PhD, M.D., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada